CLINICAL TRIAL: NCT06550401
Title: The BREAST-Q REACT: Examining the Impact of Immediate Patient-reported Outcome Feedback and Interpretation in the Perioperative Period, a Feasibility Study
Brief Title: A Study of the BREAST-Q REACT Tool for People Having Breast Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-184
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Breast Conserving Surgery; Mastectomy With Reconstruction
Keywords: BREAST-Q REACT; assessments; quality of life; 24-184

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Participants in the control group will receive the usual feedback from questionnaires completed before and after routine surgery by discussing it with their surgeon
  Interventions: Other: QuickDASH
- Intervention group (Experimental): Participants in the intervention group will receive feedback using the BREAST-Q REACT tool from questionnaires completed before and after routine surgery, in addition to the usual way by discussing it with their surgeon.
  Interventions: Other: BREAST-Q Physical Well-Being

INTERVENTIONS:
Other: BREAST-Q Physical Well-Being — This BREAST-Q domain measures pain or tightness and difficulty with mobility, such as lifting arms or running. The preoperative survey contains 10 items, whereas the postoperative survey contains 11 items. Values for BREAST-Q subscales are converted to summary scores, ranging from 0 to 100, via Q-Score software. Higher scores correlate with better patient quality of life. 37 This survey is administered as part of standard care for all patients.
  Arms: Intervention group
Other: QuickDASH — QuickDASH, also known as the Arm and Shoulder Range of Motion survey within MSK Engage is an 11-item survey that measures physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. It is currently standard of care for breast cancer surgery patients. It is a valid, reliable, and responsible survey that can be used for clinical and/or research purposes. Higher scores indicate greater disability.
  Arms: Control group

SUMMARY:
The researchers are doing this study to find out whether it is practical (feasible) to conduct a larger study looking at the effects of the BREAST-Q Real-time Engagement and Communication Tool (REACT) on people's quality of life, interactions with their doctors, and medical interventions after undergoing routine breast conserving surgery or mastectomy. The BREAST-Q REACT tool shows scores from standard questionnaires completed before and after breast surgery about overall physical wellbeing, arm pain or tightness, the ability to move the arms and perform everyday tasks, and any symptoms related to the arms, and provides feedback including recommendations and detailed information that help explain these scores and guide topics for people and their doctor to discuss.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo BCS or mastectomy followed by breast reconstruction with tissue expander, autologous tissues, or direct-to-implant, regardless of neoadjuvant chemotherapy or radiation history
* Female sex
* Able to speak and understand English
* ≥18 years of age
* Able to access the patient portal online

Exclusion Criteria:

* Patient is male
* Younger than 18 years of age
* Cannot communicate in English
* Recurrent breast cancer
* Patients without access to the internet.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast
Enrollment: 69 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
feasibility of recruitment | up to 3 months
  assessed by frequency data from initial eligibility screening to enrollment

SECONDARY OUTCOMES:
feasibility of protocol delivery | up to 3 months
  by evaluating survey completion rates and proportion of patients who are being referred to medical interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Nelson, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm